CLINICAL TRIAL: NCT04830566
Title: Effects of a Myofascial Technique on Biomechanical Properties of the Lumbar Paraspinal Muscle and Thoracolumbar Fascia in Chronic Low Back Pain Adults Assessed by Elastography, Ultrasonography and Myometry
Brief Title: Effects of a Myofascial Technique on Biomechanical Properties of the Lumbar Myofascia of Chronic Low Back Pain Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Research director, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-3572
Record Dates: First submitted 2021-03-19; First posted 2021-04-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain; Fascia properties; Thoracolumbar fascia; Myofascial release; Manual therapy; Osteopathy; Ultrasound imaging; Sonoelastography
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release technique group (Experimental)
  Interventions: Other: Myofascial release technique
- Simulated myofascial release technique group (Sham Comparator)
  Interventions: Other: Simulated Myofascial Release technique

INTERVENTIONS:
Other: Myofascial release technique — Myofascial technique on the thoracolumbar fascia and lumbar paraspinal muscles
  Arms: Myofascial release technique group
Other: Simulated Myofascial Release technique — Superficial hands contact on the lumbar area
  Arms: Simulated myofascial release technique group

SUMMARY:
Non-specific low back pain is a worldwide health issue that remains poorly understood. Some authors have shown that the thoracolumbar fascia of low back pain adults presents changes in biomechanical properties. As it is richly endowed with pain receptors, the thoracolumbar fascia could therefore be a key contributor to this chronic pain condition. Myofascial techniques (MFTs) are commonly used in manual therapy by practitioners of various backgrounds to address fascia biomechanical properties, but there is a paucity of objective evidence on their effects on tissue state. Musculoskeletal ultrasonography, sonoelastography and myometry are emerging imaging techniques that can quantify the biomechanical properties of fascia and underlying muscle. These innovative techniques could in turn contribute to a better understanding of MFTs effects on fascial properties.

The main objective of this study is to evaluate the immediate effect of a standardized MFT on the elastography features of the lumbar paraspinal muscle and fascia (i.e. myofascial unit). The secondary objectives are to evaluate the immediate effects of a MFT on: i) ultrasonography features of the myofascial unit; ii) myometry features of the myofascial unit; ii) pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years of age,
* lumbar pain and/or referred pain above or below the gluteal fold , with intensity > 3/10, persisting for > 6 months and presenting during the day > 50% of the time.

Exclusion Criteria:

* history of serious spinal or lower extremity injury or surgery in the last year
* identifiable back pain or known pathology
* known rheumatological condition
* oral or injectable corticosteroids in the lumbar spine within the last 3 months
* psychiatric disorder
* pregnancy
* manual treatment of the lumbo-sacral region 1 month prior to the experimentation and during the week of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in elastography features of the myofascial unit | Baseline (before treatment), post-treatment (immediately after treatment)
  Evaluated with a shear wave sonoelastography device.

SECONDARY OUTCOMES:
Changes in ultrasonography features of the myofascial unit | Baseline (before treatment) post-treatment (immediately after treatment)
  Evaluated with a B-mode ultrasound imaging device
Changes in myometry features of the myofascial unit | Baseline (before treatment) post-treatment (immediately after treatment)
  Evaluated with a myotonometer
Changes in pain intensity | Baseline (before treatment) post-treatment (immediately after treatment), at day 2 and at day 7 after the intervention
  Numeric rating Scale (0 to 10; minimum = 0; maximum = 10; higher score means worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Gaudreault, PhD, Study Director — Université de Sherbrooke; Mélanie Morin, PhD, Study Director — Université de Sherbrooke
Locations (1):
- Centre de recherche du Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided